CLINICAL TRIAL: NCT02015104
Title: A Randomized, Prospective, Phase II Study to Determine the Efficacy of Bacillus Calmette-Guerin (BCG) Given in Combination With PANVAC[TM] Versus BCG Given Alone in Adults With High Grade Non-Muscle Invasive Bladder Cancer (NMIBC) Who Failed at Least 1 Induction Course of BCG
Brief Title: Study of Bacillus Calmette-Guerin (BCG) Combined With PANVAC Versus BCG Alone in Adults With High Grade Non-Muscle Invasive Bladder Cancer Who Failed At Least 1 Course of BCG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Raju Chelluri, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140036; 14-C-0036
Record Dates: First submitted 2013-12-18; First posted 2013-12-19 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Bladder Cancer
Keywords: Urothelial Carcinoma; Vaccines; Immunotherapy; TICE BCG; Intravesical Treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Panvac-VF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bacillus Calmette-Guerin (BCG) + PANVAC (Experimental): Intravesical TICE BCG (50mg) once weekly starting in week 3 for a total of 6 weeks. PANVAC-V 2 x 10^8 pfu subcutaneous (SQ) at week 0 only; PANVAC-F 1 x 10^9 pfu SQ at weeks 3, 7, 11, and 15
  Interventions: Biological: BCG intravesical live (TICE Bacillus Calmette-Guerin (BCG)); Biological: PANVAC
- Bacillus Calmette-Guerin (BCG) Alone (Experimental): Intravesical TICE BCG (50mg) once weekly starting in week 3 for a total of 6 weeks
  Interventions: Biological: BCG intravesical live (TICE Bacillus Calmette-Guerin (BCG))

INTERVENTIONS:
Biological: BCG intravesical live (TICE Bacillus Calmette-Guerin (BCG)) — TICE BCG for intravesical use, is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
Biological: PANVAC — A recombinant virus vector vaccine containing genes for human carcinoembryonic antigen (CEA), mucin-1 (MUC-1) and three co-stimulatory molecules (designated Triad of costimulatory molecules (TRICOM): B7.1, intercellular adhesion molecule-1 (ICAM-1), and leukocyte function-associated antigen-3 (LFA-3).
  Arms: Bacillus Calmette-Guerin (BCG) + PANVAC

SUMMARY:
Background:

- Many cancers produce two particular proteins. The immune system can target these to attack the cancer. The PANVAC vaccine puts genes for these proteins inside a virus vaccine so the body sees the proteins as foreign invaders and attacks them. Researchers will test PANVAC on people with high grade non-muscle invasive bladder cancer. They will give it to people who have not responded to the usual treatment, bacillus Calmette-Guerin (BCG) over several weeks. They want to see if PANVAC plus BCG is better than BCG alone.

Objective:

- To compare the effects of PANVAC plus BCG therapy, to BCG therapy alone.

Eligibility:

- Adults 18 and older with high grade non-muscle invasive bladder cancer who failed at least 1 course of BCG.

Design:

* Participants will be screened with blood and urine tests and abdominal scans.
* Participants will be randomly assigned to get BCG only or BCG plus PANVAC.
* They will have up to 10 visits over 15 weeks. Most of these are part of usual cancer care.
* They will have blood and urine tests.
* All participants will get BCG in 6 weekly injections.
* One group will also get PANVAC in 5 injections over 15 weeks.
* Between weeks 17 and 20, participants will undergo tests of the tumor area as part of their usual care. They will have cystoscopy, exam under anesthesia, and bladder biopsy. Results will be used to evaluate the different treatments.
* Participants will have quarterly follow-up visits for up to 2 years.

DETAILED DESCRIPTION:
Background:

* High grade (G3) non-muscle invasive urothelial carcinoma of the bladder (stages Ta, T1, and carcinoma in situ (CIS) has a high rate of recurrence and progression
* The standard of care therapeutic agent is a single induction course of bacillus Calmette- Guerin (BCG)
* Although a second induction course can be used in patients who fail a single induction course of BCG, only 35% of patients who failed an initial induction course will experience 12 month disease-free survival after receiving a second induction course
* For those patients failing a second induction course, radical cystectomy with pelvic lymphadenectomy is the recommended treatment, although it has a high morbidity rate and a small but real mortality rate
* Therefore, there is an unmet need for localized treatment for patients who fail an initial induction course of BCG that can potentially improve upon the poor results of a second induction course of BCG
* Recently, a unique pox viral vector-based vaccine, PANVAC, has been shown to induce a cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) antigen-specific immune response against the tumor-associated antigens (TAAs), carcinoembryonic antigen (CEA) and mucin-1 (MUC-1). This vaccine also contains transgenes for three human T cell co-stimulatory molecules that can potentially augment an immune response
* We hypothesize that the combined administration of BCG and PANVAC may augment the BCG-induced cytotoxic T lymphocyte response against bladder cancer cells expressing MUC-1 and/or CEA and potentially reverse BCG failure in patients that have failed one induction course of BCG

Objectives:

-To determine if there is an improvement in disease-free survival (DFS) with BCG + PANVAC compared with BCG alone in a phase II study in non-muscle invasive high-grade urothelial carcinoma of the bladder who have failed to respond to intravesical BCG within 1 year post treatment.

Eligibility:

* Individuals who have failed at least one previous induction course of intravesical BCG, defined as histologically confirmed persistent or relapsing tumor present on post-BCG endoscopic evaluation. All BCG failures will be considered for inclusion into the study, including BCG-refractory,-resistant, and -relapsing, as defined in the Rationale and Background. For the purposes of the study, BCG-refractory and BCG-resistant subjects will be considered to have BCG-persistent disease.
* Patients who are not currently candidates for radical cystectomy (e.g. patient refuses surgery, comorbidities preclude major surgery, etc.).
* Normal organ function, Eastern Cooperative Oncology Group (ECOG) 0-2.

Design:

* This is a randomized, open label prospective, Phase II study in subjects with non-muscle invasive high grade urothelial carcinoma of the bladder who have failed at least one induction course of intravesical BCG, randomized to one of the following arms: BCG intravesical live (TICE BCG) +PANVAC or TICE BCG alone. Randomization is stratified by BCG treatment subgroup.
* All subjects will receive intravesical TICE BCG (50mg) as per usual standard of care once weekly starting in week 3 for a total of 6 weeks.
* The combination arm will receive the pox viral vaccines that contain the transgenes for CEA and MUC-1 (both with modified human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2) agonist epitopes) as well as 3 human T-cell costimulatory molecules, B7-1, intercellular adhesion molecule (ICAM-1), and lymphocyte function associated antigen 3 (LFA-3) [rV-PANVAC (vaccinia) and rFPANVAC (fowlpox)] as follows:

  * rV-PANVAC 2 x 10(8) pfu subcutaneous (SQ) at week 0 only.
  * rF-PANVAC1 x 10(9) pfu SQ at weeks 3, 7, 11, and 15.
* For this Phase II study, we will test the hypothesis that subjects in the TICE BCG +PANVAC arm have better disease-free survival than subjects in the TICE BCG alone arm.
* Patient accrual is targeted at one patient per month during the first 6 months and 1-2 patients per 1-2 months afterwards, and follow-up period after completing accrual will be 12 months post treatment.
* Based on a power of 84% and type 1 error (1-sided) of 0.15, a total of 49 subjects will need to be accrued.
* Allowing for a proportion of the subjects not being evaluable, a maximum of 54 subjects will be accrued.

ELIGIBILITY:
* INCLUSION CRITERIA:

3.1.1.1 Patients must have histologically confirmed localized high grade (G3) transitional cell carcinoma (urothelial carcinoma) of the bladder that is stage Ta, T1, and/or carcinoma in-situ (CIS) confirmed by the Laboratory of Pathology, National Cancer Institute (NCI) 45 days prior to study entry. This can be obtained at an outside hospital prior to entry into the study or at the NCI. However, all outside pathology specimens will require that the formalin-fixed paraffin embedded tissues be re-read by the Laboratory of Pathology, NCI. For patients enrolled at collaborating trial sites, diagnosis must be confirmed by the Department of Pathology at the institution where the patient is enrolled on the trial.

Pathology can also be reviewed by the Laboratory of Pathology at the NCI if the participating trial site prefers another pathologic evaluation.

3.1.1.2 Patients have failed at least one previous induction course of intravesical Bacillus Calmette-Guerin (BCG), defined as histologically confirmed persistent or relapsing tumor present on post-BCG endoscopic evaluation. All BCG failures will be considered for inclusion into the study, including BCG-refractory, -resistant, and relapsing, as defined in the Rationale and Background. For the purposes of the study, BCG-refractory and BCG-resistant subjects will be considered to have BCG-persistent disease.

3.1.1.3 Patients who are not currently candidates for radical cystectomy (e.g. patient refuses surgery, comorbidities preclude major surgery, etc.).

3.1.1.4 Age >18 years.

--Because no dosing or adverse event data are currently available on the use of BCG in combination with PANVAC in patients <18 years of age, children are excluded from this study.

3.1.1.5 Eastern Cooperative Oncology Group (ECOG) performance status <2.

3.1.1.6 Patients must have normal organ and marrow function as defined below:

* absolute neutrophil count greater than or equal to1,500/mcL
* platelets greater than or equal to 50,000/mcL
* total bilirubin less than or equal to 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 X institutional upper limit of normal
* estimated glomerular filtration rate (GFR) (calculated using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation) greater than or equal to 30 mL/min/1.73 sq.m.

3.1.1.7 Computerized Tomography (CT) urogram or Magnetic Resonance Imaging (MRI) urogram. If urogram protocol not available or contrast allergy/poor renal function preclude such imaging, then noncontrast CT or MRI of the abdomen/pelvis within 45 days of study entry will suffice.

3.1.1.8 Chest x-ray negative for metastatic disease.

3.1.1.9 Ability of patient to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

3.1.2.1 Previous pelvic radiation for bladder or prostate cancer if performed <12 months prior to enrollment into the study.

3.1.2.2 Patients who are receiving any other concurrent investigational agents (patients are eligible to enroll 4 weeks after completion of prior agent).

3.1.2.3 Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. There will be at least a 3 week delay from the time of a previous bladder biopsy/transurethral resection of bladder tumor (TURBT) to allow for adequate bladder healing prior to enrollment.

3.1.2.4 Patients with a history of encephalitis, multiple sclerosis, or seizures within the last year (from seizure disorder or brain metastasis) should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

3.1.2.5 History of allergy or untoward reaction to prior vaccination with vaccinia virus

3.1.2.6 Patients should have no evidence of being immunocompromised as listed below:

* Human immunodeficiency virus positivity due to the potential for decreased tolerance and risk for severe side effects
* Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity. Patients with endocrine disease that is controlled by replacement therapy including thyroid disease and adrenal disease and vitiligo may be enrolled.
* History of splenectomy

3.1.2.7 Uncontrolled intercurrent illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, active second malignancy other than a cancer that has been successfully treated resulting in a high likelihood of long-term survival (e.g. completely resected basal cell or squamous cell carcinoma of the skin, stage 1 renal cell carcinoma treated with partial nephrectomy, treated low risk prostate cancer, etc.), inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis), active diverticulitis, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

3.1.2.8 Pregnant women are excluded from this study because the vaccines used in the study may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the vaccine, breastfeeding should be discontinued if the mother is treated with vaccines. These potential risks may also apply to other agents used in this study. Patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately

3.1.2.9 Concurrent use of systemic steroids, except for physiologic doses of systemic steroids for replacement or local (topical, nasal, or inhaled) steroid use. Limited doses of systemic steroids to prevent intravenous (IV) contrast, allergic reaction, or anaphylaxis (in patients who have known contrast allergies) are allowed. Although topical steroids are allowed, steroid eye-drops are contraindicated

3.1.2.10 Altered immune function, including immunodeficiency or history of immunodeficiency; eczema; history of eczema, or other eczematoid skin disorders; or those with acute, chronic or exfoliative skin conditions (e.g. atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds). There is an increased risk to patients or contacts with eczema, atopic dermatis, and other immune deficiencies who are at risk for eczema vaccination.

3.1.2.11 Medical conditions which, in the opinion of the investigators, would jeopardize the patient or the integrity of the data obtained

3.1.2.12 Serious hypersensitivity reaction to egg products

3.1.2.13 Chronic hepatitis infection, including B and C, because of potential immune impairment

3.1.2.14 Clinically significant cardiomyopathy or cardiac complications, including recent myocardial infarction or cerebrovascular accident within one year, and/or unstable or uncontrolled angina

3.1.2.15 Previous intolerance to BCG intravesical therapy suggested by development of systemic BCG infection in the past and/or grade 4 or greater adverse effect by Common Terminology Criteria in Adverse Events (CTCAE) v4.0.

3.1.2.16 Patients unable to avoid close contact or household contact with the following high-risk individuals for three weeks after the Day 1 vaccination: (a) children less than or equal to 3 years of age, (b) pregnant or nursing women, (c) individuals with prior or concurrent extensive eczema or other eczematoid skin disorders, or (d) immunocompromised individuals, such as those with human immunodeficiency virus (HIV).

3.1.3 Inclusion of Women and Minorities:

Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raju Chelluri, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulley JL, Arlen PM, Tsang KY, Yokokawa J, Palena C, Poole DJ, Remondo C, Cereda V, Jones JL, Pazdur MP, Higgins JP, Hodge JW, Steinberg SM, Kotz H, Dahut WL, Schlom J. Pilot study of vaccination with recombinant CEA-MUC-1-TRICOM poxviral-based vaccines in patients with metastatic carcinoma. Clin Cancer Res. 2008 May 15;14(10):3060-9. doi: 10.1158/1078-0432.CCR-08-0126. PMID 18483372
- [Background] Kavoussi LR, Torrence RJ, Gillen DP, Hudson MA, Haaff EO, Dresner SM, Ratliff TL, Catalona WJ. Results of 6 weekly intravesical bacillus Calmette-Guerin instillations on the treatment of superficial bladder tumors. J Urol. 1988 May;139(5):935-40. doi: 10.1016/s0022-5347(17)42722-4. PMID 3361667
- [Background] Crawford ED. Intravesical therapy for superficial cancer: need for more options. J Clin Oncol. 2002 Aug 1;20(15):3185-6. doi: 10.1200/JCO.2002.20.15.3185. No abstract available. PMID 12149286
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0036.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacillus Calmette-Guerin (BCG) + PANVAC: Intravesical TICE BCG (50mg) once weekly starting in week 3 for a total of 6 weeks. PANVAC-V 2 x 10^8 pfu subcutaneous (SQ) at week 0 only; PANVAC-F 1 x 10^9 pfu SQ at weeks 3, 7, 11, and 15
  TICE Bacillus Calmette-Guerin (BCG): TICE BCG for intravesical use, is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
  PANVAC: A recombinant virus vector vaccine containing genes for human carcinoembryonic antigen (CEA), mucin-1 (MUC-1) and three co-stimulatory molecules (designated Triad of costimulatory molecules (TRICOM): B7.1, intercellular adhesion molecule-1 (ICAM-1), and leukocyte function-associated antigen-3 (LFA-3).
- Bacillus Calmette-Guerin (BCG) Alone: Intravesical TICE BCG (50mg) once weekly starting in week 3 for a total of 6 weeks
  TICE Bacillus Calmette-Guerin (BCG): TICE BCG for intravesical use, is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
Period: Overall Study
Arm/Group | Bacillus Calmette-Guerin (BCG) + PANVAC | Bacillus Calmette-Guerin (BCG) Alone
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Withdrew consent after first dose drug | 1 | 0
Not completed — Withdrew consent prior to treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bacillus Calmette-Guerin (BCG) + PANVAC: Intravesical TICE BCG (50mg) once weekly starting in week 3 for a total of 6 weeks. PANVAC-V 2 x 10^8 pfu subcutaneous (SQ) at week 0 only; PANVAC-F 1 x 10^9 pfu SQ at weeks 3, 7, 11, and 15
  TICE Bacillus Calmette-Guerin (BCG): TICE BCG for intravesical use, is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
  PANVAC:A recombinant virus vector vaccine containing genes for human carcinoembryonic antigen (CEA), mucin-1 (MUC-1) and three co-stimulatory molecules (designated Triad of costimulatory molecules (TRICOM): B7.1, intercellular adhesion molecule-1 (ICAM-1), and leukocyte function-associated antigen-3 (LFA-3).
- Total: Total of all reporting groups
Arm/Group | Bacillus Calmette-Guerin (BCG) + PANVAC | Bacillus Calmette-Guerin (BCG) Alone | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.73 (11.21) | 72.66 (9.61) | 71.7 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32
Enrollment Disease Status [Count of Participants; unit: Participants] — TNM Classification in non-muscle invasive bladder cancer: Ta - Non-invasive papillary carcinoma; T1 - Tumor invades the subepithelial connective tissue.
  CIS - Carcinoma in-situ
  Participants
    CIS | 3 | 3 | 6
    Ta + CIS | 2 | 0 | 2
    T1 + CIS | 0 | 1 | 1
    Ta | 8 | 7 | 15
    T1 | 3 | 4 | 7
    Unknown | 0 | 1 | 1
Number of Patients with≥2 Prior Bacillus Calmette-Guerin (BCG) Induction Before Treatment [Count of Participants; unit: Participants] | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Recurrence (Recurrence-free Survival (RFS)) With Bacillus Calmette-Guerin (BCG) + PANVAC Compared With BCG Alone at 6 and 12 Months
Description: RFS is defined as the time from the start of intravesical Bacillus Calmette-Guerin (TICE BCG) therapy (week 3) until disease recurrence or death due to any cause in each arm. Recurrence is suspected and/or determined by urine cytology and/or cystoscopic exam and then confirmed pathologically after a transurethral resection of bladder tumor (TURBT). Positive cytology in the absence of pathologic confirmation is not considered to be a recurrence.
Time Frame: Assessed from start of therapy to 6 and 12 months following therapy
Population: One patient withdrew consent after the first dose of drug in the BCG + PANVAC group. One patient withdrew consent prior to treatment in the BCG Alone group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bacillus Calmette-Guerin (BCG) + PANVAC | Bacillus Calmette-Guerin (BCG) Alone
Number analyzed (Participants) | 15 | 15
percentage of participants
  6 months | 66 [46.6 to 95.3] | 60 [39.5 to 90.7]
  12 months | 44.4 [24.8 to 79.7] | 42.9 [22.9 to 80.0]

2. Secondary Outcome: Percentage of Participants Without Progression (Progression-Free Survival (PFS)) at 6 and 12 Months
Description: PFS is the duration of time from start of TICE BCG therapy (week 3) to time of progression or death due to any cause in each study arm, whichever occurs first. Progression is defined as upstaging from a lower stage to a higher stage (e.g., Ta to T1 or T1 to T2-4; or any N+ or M+ in these high grade tumors.).TNM Classification in non-muscle invasive bladder cancer: Ta = Non-invasive papillary carcinoma; T1 = Tumor invades the subepithelial connective tissue; T2-4 = size of primary tumor; N+ or M+ = lymph node involvement and metastasis.
Time Frame: Assessed from start of therapy to 6 and 12 months following therapy
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bacillus Calmette-Guerin (BCG) + PANVAC | Bacillus Calmette-Guerin (BCG) Alone
Number analyzed (Participants) | 15 | 15
percentage of participants
  6 months | 79 [59.8 to 100] | 93 [80.3 to 100]
  12 months | 78.5 [59.8 to 100] | 79.6 [56.9 to 100]

3. Secondary Outcome: Time to Recurrence
Description: TTR is the duration of time measured from the start of TICE BCG therapy (week 3) until recurrence is noted. Recurrence is suspected and/or determined by urine cytology and/or cystoscopic exam and then confirmed pathologically after a TURBT. Positive cytology in the absence of pathologic confirmation is not considered to be a recurrence.
Time Frame: Week 3 until recurrence or 12 months (whichever occurred first)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bacillus Calmette-Guerin (BCG) + PANVAC | Bacillus Calmette-Guerin (BCG) Alone
Number analyzed (Participants) | 15 | 15
Months | 9.9 [3.7 to NA] — The calculation of the confidence intervals is based on the number of occurrences (events). The upper limit of confidence interval cannot be calculated. This is probably due to the small sample size and number of events in each arm. | 11.7 [4 to NA] — The calculation of the confidence intervals is based on the number of occurrences (events). The upper limit of confidence interval cannot be calculated. This is probably due to the small sample size and number of events in each arm.

4. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Serious and non-serious adverse events were assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events were assessed from the date treatment consent was signed to the date off study. Approximately 50 months and 12 days for BCG + PANVAC Arm/Group, and 43 months and 12 days for BCG Alone Arm/Group.
Population: One patient withdrew consent prior to treatment in the BCG Alone group.
Measure: Count of Participants; unit: Participants
Arm/Group | Bacillus Calmette-Guerin (BCG) + PANVAC | Bacillus Calmette-Guerin (BCG) Alone
Number analyzed (Participants) | 16 | 15
Participants | 16 | 13

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from treatment start date until date of death or date last known alive.
Time Frame: up to 50 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- BCG + PANVAC: Intravesical TICE BCG (50mg) once weekly starting in week 3 for a total of 6 weeks. PANVAC-V 2 x 10^8 pfu subcutaneous (SQ) at week 0 only; PANVAC-F 1 x 10^9 pfu SQ at weeks 3, 7, 11, and 15
  TICE Bacillus Calmette-Guerin (BCG): TICE BCG for intravesical use, is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
  PANVAC: A recombinant virus vector vaccine containing genes for human carcinoembryonic antigen (CEA), mucin-1 (MUC-1) and three co-stimulatory molecules (designated Triad of costimulatory molecules (TRICOM): B7.1, intercellular adhesion molecule-1 (ICAM-1), and leukocyte function-associated antigen-3 (LFA-3).
- BCG Alone: Intravesical TICE BCG (50mg) once weekly starting in week 3 for a total of 6 weeks
  TICE Bacillus Calmette-Guerin (BCG): TICE BCG for intravesical use, is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis
Arm/Group | BCG + PANVAC | BCG Alone
Number analyzed (Participants) | 15 | 15
Months | 41.4 [22.6 to NA] — Due to few deaths the upper 95% confidence limit is not reached for the BCG+PANVAC arm. | 35.1 [0 to NA] — Due to few deaths the upper 95% confidence limit is not reached for the BCG alone arm.

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date treatment consent was signed to the date off study. Approximately 50 months and 12 days for BCG + PANVAC, and 43 months and 12 days for BCG Alone.
Description: One patient withdrew consent prior to treatment in BCG Alone group.
Arm/Group | BCG + PANVAC | BCG Alone
All-Cause Mortality (participants affected / at risk) | 3/15 | 2/15
Serious Adverse Events (participants affected / at risk) | 3/15 | 3/15
Other Adverse Events (participants affected / at risk) | 15/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG + PANVAC (N=15) | BCG Alone (N=15)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Death, NOS (General disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG + PANVAC (N=15) | BCG Alone (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 6 (7) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (9) | 5 (8)
Fever (General disorders) | 4 (5) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 3 (9) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 5 (12) | 5 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 12 (20) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (3) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (9) | 3 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, 3+ Glucose in urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (4) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (2) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (3) | 5 (13)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (6)
Urinary retention (Renal and urinary disorders) | 1 (1) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (6) | 5 (12)
Urinary urgency (Renal and urinary disorders) | 4 (4) | 3 (7)
Urine discoloration (Renal and urinary disorders) | 3 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 2 (2) | 3 (7)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, fecal urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (7)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Head cold
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Red blotch on forearm
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT02015104/Prot_SAP_002.pdf
  • Informed Consent Form (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT02015104/ICF_001.pdf